CLINICAL TRIAL: NCT02739724
Title: Comparison Between Classic and Single Port Access Laparoscopy for Adnexal Surgery on Postoperative Pain: a Randomized Study.
Brief Title: Benefits of Laparoscopy by Single Port Access for Adnexal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A01217-42; 2015-32 (Other: AP-HM)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Adnexal Pathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classic laparoscopy (Active Comparator): Patients will undergo laparoscopy surgery with classic laparoscopy technic.
  Interventions: Procedure: Adnexal surgery
- Laparoscopy single port access (Experimental): Patients will undergo laparoscopy surgery by single port access technic.
  Interventions: Procedure: Adnexal surgery

INTERVENTIONS:
Procedure: Adnexal surgery

SUMMARY:
Introduction

Single port access (SPA) is a recent laparoscopic technic evaluated in several pathologies. Benefits of this technic is poorly reported concerning adnexal surgical procedures. Results of both randomised studies including adnexectomy and ovarian cystectomy are discordants. So it seems interesting to conduct a new study about this technic. Aim of this study is to compare postoperative pain after laparoscopic surgery for adnexal pathology by SPA or classic laparoscopy (CL).

Materiel and Methods

We purpose a monocentric-randomised study. Inclusion criteria are women over 18 years requiring laparoscopic surgery for adnexal pathology with stratification for procedure (adnexectomy or ovarian cystectomy). After informed consent, patients will be randomised in two groups: laparoscopy with SPA and laparoscopy with CL. The main objective is postoperative pain evaluation at 24 hours. Secondary objectives are characteristics and perioperative complications, duration of procedure, postoperative quality of life and immediate postoperative pain.

We hypothesis laparoscopy with SPA reduces postoperative pain at 24 hours of 2 pts (analogic scale 0-10). The estimated size of population number is 54 per group and 108 for the study.

Expected results

We expected a significant decrease of postoperative pain with SPA technic. This data will be interesting to promote use of SPA technic for adnexal surgery.

ELIGIBILITY:
Inclusion Criteria:

Presumed benign adnexal disease Adnexal pathologies treated between 7:00 AM and 10:00 PM Signed informed consent Patient presenting no contraindication to laparoscopy

Exclusion Criteria:

Salpingitis and twist annexes. The patient does not fluently read French.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measured with visual analog scale | Postoperative pain evaluation at 24 hours

SECONDARY OUTCOMES:
Postoperative pain measured with visual analog scale | 2 hours, 4 hours, 6 hours, 1 month
timing in minutes between incision and suture | 4 hours
Blood lost in milliliters (mls) | 1 hour
Inpatient numbers of days | 1 month
Non steroid anti inflammatory numbers of pills taken | 1 month
number of convertion to laparotomy, Postoperative hernia | 1 month
visual analog scale for cosmetic satisfaction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — AP-HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmitt A, Crochet P, Baumstark K, Tourette C, Poizac S, Pivano A, Boubli L, Cravello L, Agostini A. Effect of laparoscopy by single-port endoscopic access in benign adnexal surgery: study protocol for a randomized controlled trial. Trials. 2018 Jan 15;19(1):38. doi: 10.1186/s13063-017-2429-y. PMID 29335017